CLINICAL TRIAL: NCT02264509
Title: Prevalence and Risk Factors of Arterial Insufficiency in Patients With HIV / AIDS
Brief Title: Peripheral Arterial Insufficiency Associated With HIV/AIDS
Acronym: AIHIV
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Carlos Hinojosa, subdirector of clinical research, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: InstitutoNCMNSZ-CIIBH693
Record Dates: First submitted 2014-09-12; First posted 2014-10-15 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Arterial Insufficiency; Acquired Immunodeficiency Syndrome; HIV
Keywords: Arterial Insufficiency; Human Immunodeficiency Virus; Atherosclerosis; Ankle-brachial index; HAART
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arterial insufficiency and HIV: Of a cohort of 206 HIV patients will be randomly selected 206 for Ankle-brachial index to identify wich suffer symptomatic or asymptomatic arterial insufficiency
  Interventions: Procedure: Ankle-Brachial index

INTERVENTIONS:
Procedure: Ankle-Brachial index — The only procedure to be performed is the measurement of ABI for the diagnosis of arterial insufficiency.

SUMMARY:
The purpose of this study is to determine the risk factors associated with the occurrence of arterial insufficiency in patients with HIV / AIDS, and to identify the prevalence of this disease. The estimated prevalence is 10%, similar to that reported in the general population.

DETAILED DESCRIPTION:
A case study nested in a cohort of patients with HIV / AIDS at Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico, with a cohort of 1500 patients , a sample size of 206 individuals was calculated. Data collection was performed in a prospective cross shape.

During the interview, written informed consent for inclusion in the study, along with a standard query of vascular surgery in which the patient's history as well as cardiovascular risk factors. Also, a vascular physical examination including palpation of pulses in upper and lower extremities (brachial, radial, ulnar, femoral, popliteal, posterior tibial and dorsalis pedis), femoral murmurs search and determining ankle / brachial indexes with a standardized method.

In determining the ABI was counted with a Doppler ultrasound 8 mHz, transducer gel and a sleeve for manual measurement of blood pressure, 20% longer than the largest diameter of the arm circumference.

If the patient is diagnosed with, symptomatic or asymptomatic arterial insufficiency, ABI measurements were performed at rest and effort, plus pressure index finger-arm or plethysmography. Patients with altered rates were followed in vascular surgery care.

The data were recorded in a single database unique protected by password. The results were analyzed using the statistical program STATA v 9.0.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HIV / AIDS are included in active consultation of Infectious Diseases INCMNSZ and sign informed consent.

Exclusion Criteria:

* Patients who do not wish to participate in the study and those who did not complete their interview and vascular physical examination.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The 206 patients will be randomly selected from the cohort HIV / AIDS INCMNSZ, which have confirmed diagnosis of the disease and wish to participate in the study, without a disease that put life in imminent danger.
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Arterial insufficiency | 1 time
  Arterial insufficiency is measured by Ankle / brachial index described as ABI<0.9 or ABI >1.2

SECONDARY OUTCOMES:
Gender | 1 time
  Male or Female
Age | 1 time
  Number of years
Diabetes mellitus | 1 time
  Defined as diagnosis in previous notes in the file or use of oral hypoglycemic agents.
Hypercholesterolemia | 1 time
  Defined as the last digit of C-LDL in serum of the patient, which is more than 150 mg / dL.
Hypertriglyceridemia | 1 time
  Defined as the last digit of the patient's serum triglycerides, which is greater than 200 mg / dL.
Hypoalphalipoproteinemia | 1 time
  Defined as the last digit of HDL-C in patient serum, which is less than 50 mg / dL.
Hypertension (High blood pressure) | 1 time
  Defined as diagnosis in previous notes or use of antihypertensives.
Ischemic heart disease | 1 time
  Defined as previous heart attack.
Stroke | 1 time
  Defined as previous diagnosis in the record.
Smoking | 1 time
  Smoking yes or no.
Smoking index | 1 time
  Smoking index defined as the number of cigarettes smoked per day by the number of years of smoking divided by 20.
Drug abuse | 1 time
  Defined as use or history of use of drugs of abuse investigated during the interview
AIDS | 1 time
  Defined as confirmatory serologic diagnosis of HIV associated with AIDS-defining illnesses
Diagnostic Time of HIV | 1 time
  Defined as the time interval in months from diagnosis of HIV to interview for the research protocol.
Viral Load | 1 time
  Defined as the last number of copies of certain virus in patient serum in the record.
CD4 | 1 time
  Defined as the final determination of number of CD4 in serum.
HAART (Highly active anti-retroviral therapy) | 1 time
  Defined as use of at least one drug with anti-retroviral activity.
Time HAART | 1 TIME
  Defined as a period in months

OTHER OUTCOMES:
HIV | 1 time
  Defined as confirmatory serological diagnosis of HIV (ELISA + Western Blot)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A. Hinojosa, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Ana Elsa Núñez Salgado, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Laura Jael del C. Ortiz López, MD, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Jaime Omar Herrera Cáceres, MD, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Brenda E. Crabtree Ramirez, MD, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Juan Sierra Madero, MD, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, D.f., Mexico, Mexico

REFERENCES:
- [Derived] Hinojosa CA, Nunez-Salgado AE, Anaya-Ayala JE, Laparra-Escareno H, Ortiz-Lopez LJ, Herrera-Caceres JO, Crabtree-Ramirez BE, Sierra-Madero JG. Prevalence and variables associated with an abnormal ankle-brachial index among patients with human immunodeficiency virus/acquired immunodeficiency syndrome. Vascular. 2018 Oct;26(5):540-546. doi: 10.1177/1708538118770542. Epub 2018 Apr 13. PMID 29649953